CLINICAL TRIAL: NCT04658914
Title: Human Challenge With Live-attenuated Rotavirus to Assess Next-generation Rotavirus Vaccines in Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Medical Research Council (Other Government); PATH (Other); University of Liverpool (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRC Rotavirus HIC
Record Dates: First submitted 2020-11-18; First posted 2020-12-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Diarrhea; Diarrhea Rotavirus
Keywords: Human Infection Challenge
MeSH Terms: conditions — Diarrhea | interventions — RIX4414 vaccine

STUDY DESIGN:
Intervention Model Description: single centre open label study, randomized, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- rotarix only (No Intervention): Rotarix will be administered at 6 and 10 weeks of age following the national Expanded Program for Immunization (EPI) schedule. A challenge dose of Rotarix will be administered at 18 weeks of age and stool samples collected just before challenge and 5, 7 & 9 days later.
- P2 VP8 only (Experimental): Parenteral P2-VP8 subunit vaccine will be administered at 6, 10 and 14 weeks of age. A challenge dose of Rotarix will be administered at 18 weeks of age and stool samples collected just before challenge and 5, 7 & 9 days later.
  Interventions: Biological: Trivalent P2-VP8
- Rotarix + 1 dose P2-VP8 (Experimental): Rotarix will be administered at 6 and 10 weeks of age, followed by parenteral P2-VP8 subunit vaccine at 14 weeks of age. A challenge dose of Rotarix will be administered at 18 weeks of age and stool samples collected just before challenge and 5, 7 & 9 days later.
  Interventions: Biological: Rotarix; Biological: Trivalent P2-VP8
- Rotarix + 3 doses P2-VP8 (Experimental): Rotarix and parenteral P2-VP8 subunit vaccine will be coadministered at 6 and 10 weeks of age, with an additional dose of P2-VP8 subunit vaccine administered at 14 weeks of age. A challenge dose of Rotarix will be administered at 18 weeks of age and stool samples collected just before challenge and 5, 7 & 9 days later.
  Interventions: Biological: Rotarix; Biological: Trivalent P2-VP8

INTERVENTIONS:
Biological: Rotarix — Live-attenuated oral human rotavirus vaccine (Rotarix) manufactured by GlaxoSmithKline containing at least 10^6 CCID50(median cell culture infective doses) of G1P[8] rotavirus, RIX4414 strain produced in Vero cells. This vaccine is an oral suspension with a single dose (1.5ml) administered using an oral applicator.
  Arms: Rotarix + 1 dose P2-VP8; Rotarix + 3 doses P2-VP8
Biological: Trivalent P2-VP8 — Trivalent P2-VP8 subunit vaccine manufactured by SK Chemicals containing 90ug of each VP8 antigen derived from P[4] (DS-1), P[6] (1076), and P[8] (Wa) rotavirus strains fused to the P2 epitope from tetanus toxoid and adsorbed to aluminium hydroxide. A single dose (0.5ml) of this vaccine is administered intramuscularly through injection.
  Arms: P2 VP8 only; Rotarix + 1 dose P2-VP8; Rotarix + 3 doses P2-VP8

SUMMARY:
Despite the widespread introduction of vaccines against Rotavirus, Rotavirus continues to be a cause of significant morbidity and mortality in the developing world. This study will assess protection against rotavirus infection and investigate immune correlates of protection following vaccination with a novel trivalent VP8 subunit rotavirus vaccine used alone or in combination with oral rotavirus vaccine.

DETAILED DESCRIPTION:
This is a randomized, open-label clinical trial of Rotarix and trivalent VP8 subunit vaccine given alone or in combined schedules to 720 infants in Zambia at 6, 10 and 14 weeks followed by challenge at 18 weeks used to assess mucosal immunity.

Potential participants will be identified through antenatal and child health monitoring clinics in selected facilities in Lusaka Zambia. Interested parents will be invited to the clinical research site for informed consent procedures and assessment of eligibility. Children meeting the eligibility criteria with written informed consent for participation will be randomized to one of the four available study arms using simple randomization in block sizes of 8. Blood, stool, and saliva samples will be collected prior to completing vaccination according to randomization arm. All parents/guardians will be provided with post immunisation diary cards to document any reactions following vaccination. Trained study staff will contact parents and guardians of enrolled participants weekly to enquire on the child's health and assist with documentation of solicited reactions following vaccinations.

Enrolled children will be followed up for at least five months following enrollment. Follow up vaccinations will be provided each month until all children have completed all assigned study vaccinations. Upon completion of study vaccination, participants will be challenged with oral rotavirus vaccine, Rotarix TM to assess mucosal immunity.

Primary outcome:

The primary objective of the study will be to detect a reduction in the proportion of children shedding vaccine rotavirus in stool at any timepoint 5-9 days after challenge, among children immunized with P2-VP8 subunit vaccine alone or in combination with Rotarix, compared with infants receiving Rotarix alone. The primary outcomes will be prevalence of rotavirus (Rotarix) shedding at any timepoint in samples collected 5,7 and 9 days after challenge.

Secondary outcomes:

i.) Seroconversion following vaccination: Detection of an increase in seroconversion in either of the combined vaccination arms compared with Rotarix alone.

ii.) Immune boosting. We will compare the number of gut-homing (alpha 4 beta 7+) Immunoglobulin A (IgA) and Immunoglobulin G (IgG) rotavirus VP8-specific Antibody secreting cells (ASCs) 7 days after the third clinic visit in 50 infants from each study arm (i.e. after the first VP8 vaccine booster dose, after the third VP8 vaccine dose (alone or in combination with Rotarix), or after no vaccine (control) in the Rotarix only arm).

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants as established by medical history and physical examination.
* Infants will be 6-10 weeks old at time of enrollment
* parents plan to remain in the area for the duration of the study.
* Parent/guardian understands the study procedures and willing to provide informed consent to participate in the study

Exclusion Criteria:

* Acutely unwell
* Infant or infant's mother has syndromic or documented evidence of being immunocompromised (independent of HIV status)
* Known allergy to any vaccine component
* Previously received rotavirus vaccine
* Received immunosuppressive medication
* Major congenital or genetic abnormality
* Any condition in the parents/infant that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give informed consent.
* Participant's parents not available or willing to accept active follow-up by the study staff

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Vaccine Shedding | 5-9 days after Challenge
  to detect a reduction in the proportion of children shedding vaccine rotavirus in stool at any timepoint 5 -9 days after challenge, among children immunized with P2-VP8 subunit vaccine alone or in combination with Rotarix, compared with infants receiving Rotarix alone. We estimate that approximately 50% (range 30-70%) of children previously vaccinated with 2 doses of Rotarix will shed Rotarix detected by Polymerase Chain Reaction (PCR) at any timepoint 5-9 days after challenge

SECONDARY OUTCOMES:
Seroconversion following vaccination | 14 and 18 weeks of age
  Seroconversion After 2 doses of Rotarix in Zambia seroconversion was 60% (130/216) in an earlier study and 45% (10/22) in our Medical Research Council UK MRC-funded pilot of Rotarix challenge, based on IgA to whole virus cell culture lysate (largely anti -VP6 antibodies). Seroconversion based on anti-VP8 antibodies has not been studied after Rotarix administration but may be similar.
Immune boosting | 7 days after 3rd clinic visit
  i.) We will compare the number of gut-homing (alpha 4 beta 7+) IgA and IgG rotavirus VP8-specific ASCs 7 days after the third clinic visit in 50 infants from each study arm (i.e. after the first VP8 vaccine booster dose, after the third VP8 vaccine dose (alone or in combination with Rotarix), or after no vaccine (control) in the Rotarix only arm).

CONTACTS AND LOCATIONS:
Overall Officials: Roma Chilengi, MD, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- Chawama first level hospital, Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Communicate with the participants results of the study and plans to share de-identified data. Disseminate to internal research meetings as well as the Ministry of Health Zambia.
  Submit manuscripts, publications, in peer review journal and also present at local and international scientific conferences
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after study completion